CLINICAL TRIAL: NCT03132389
Title: Prevalence of Sexually Transmitted Infections Among People Attending the Sexual Assault Centre in Oslo, Norway: a Cohort Study at the Sexual Assault Centre in Oslo, Norway.
Brief Title: Prevalence of Sexually Transmitted Infections Among People Attending the Sexual Assault Centre in Oslo, Norway.
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Odd Martin Vallersnes, Associate professor, University of Oslo
Other Study IDs: 2016/2279/REK
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Sexual Assault and Rape; Sexually Transmitted Diseases
Keywords: Sexual assault; Sexually transmitted diseases; Chlamydia trachomatis; Mycoplasma genitalium; Neisseria gonorrhoeae; Hepatitis B and C; HIV; Syphilis; Follow up visits after sexual assault
MeSH Terms: conditions — Sexually Transmitted Diseases; Hepatitis B; Syphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients attending after a sexual assault: Patients attending and examined after sexual assault at the Sexual Assault Centre in Oslo, who have given informed consent to inclusion in the study.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — All patients included in the study will be offered the same examination and treatment procedure as the patients who are not included. Identical procedures and examinations will be performed in participants and non-participants.

SUMMARY:
In this study the investigators seek to register the prevalence of sexually transmitted infections (STI) among people attending the Sexual Assault Centre in Oslo, Norway. The main aim of this study is to gather representative data on STIs after sexual assaults. Consequently, if the attendance for medical follow up turns out to be good/sufficient, prophylactic (antibiotic) treatment can potentially be omitted.

DETAILED DESCRIPTION:
Patients who attend sexual assault centres are often concerned about being infected with STIs. Therefore, the patients attending sexual assault centres are offered examination and often receive prophylactic treatment against some STIs (e.g. chlamydia trachomatis, HIV and hepatitis B).

In this study, the investigators seek to register the prevalence of STI among people attending the Sexual Assault Centre in Oslo, Norway. The primary aim of the study is to gather representative data on STIs after a sexual assault. Furthermore, the investigators want to evaluate if there are any variables that can predict transmission after a sexual assult. Results from this study will also be compared with findings of STI in the general population.

At the Sexual Assault Centre in Oslo, Norway, patients are routinely offered three medical follow up consultations. Consequently, if the attendance at follow up visits turns out to be adequate, prophylactic (antibiotic) treatment can potentially be omitted.

Since victims of assault are in a vulnerable situation, it would be useful to be able to inform them more precisely about infection risk and provide adequate prophylactic treatment. More knowledge about the incidence of infection after abuse will increase patient safety and improve the quality of treatment for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending and examined after sexual assault at the Sexual Assault Centre in Oslo (at Oslo Accident and Emergency Outpatient Clinic).
* Written informed consent

Exclusion Criteria:

* Patients who only had a consultation only with a social worker and no medical examination.
* Unable to communicate in Norwegian, Swedish, Danish or English language

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending and examined after sexual assault at the Sexual Assault Centre in Oslo (at Oslo Accident and Emergency Outpatient Clinic).
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Results of the STI-tests taken at the primary examination and at follow up. | 1 week
  Results of the STI-tests (i.e. Chlamydia trachomatis, Mycoplasma genitalium, Neisseria gonorrhoeae, Hepatitis B, Hepatitis C, HIV, Syphilis) taken at the primary attendance and at follow up.

SECONDARY OUTCOMES:
Attendance percentage for follow up visits. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mette Brekke, Professor, Study Director — University of Oslo
Locations (1):
- Sexual Assault Centre in Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skjaelaaen K, Nesvold H, Brekke M, Sare M, Landaas ET, Mdala I, Olsen AO, Vallersnes OM. Sexually transmitted infections among patients attending a sexual assault centre: a cohort study from Oslo, Norway. BMJ Open. 2022 Dec 1;12(12):e064934. doi: 10.1136/bmjopen-2022-064934. PMID 36456026